CLINICAL TRIAL: NCT03822910
Title: Hippocampal Memory Circuits in Delusions
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-00656
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Matched Healthy Controls
  Interventions: Diagnostic Test: Pattern Separation Paradigm; Diagnostic Test: Sequential Associative Mismatch Paradigm; Diagnostic Test: Encoding Plasticity Paradigm
- Firt Episode Psychosis (FEP): subjects before and after antipsychotic treatment
  Interventions: Diagnostic Test: Pattern Separation Paradigm; Diagnostic Test: Sequential Associative Mismatch Paradigm; Diagnostic Test: Encoding Plasticity Paradigm

INTERVENTIONS:
Diagnostic Test: Pattern Separation Paradigm — Will be used to investigate dentate gyrus (DG) and hippocampal CA3 subfield as reflected by the difference in brain activation in response to same as previously seen (OLD) vs similar to previously seen (SIM) objects in first episode (FEP) subjects before and after treatment.
Diagnostic Test: Sequential Associative Mismatch Paradigm — used to reflect activation of CA1 in response to mismatching information compared to memory of the stimulus in FEP subjects before and after antipsychotic treatment and in matched Healthy Control (HC).
Diagnostic Test: Encoding Plasticity Paradigm — Used to evaluate plasticity of hippocampal Intrinsic Functional Connectivity (IFC) in response to memory consolidation in FEP subjects before and after antipsychotic treatment and in matched HC.

SUMMARY:
This study will investigate dentate gyrus (DG) and hippocampal CA3 sub field function, using the pattern separation paradigm, as reflected by the difference in brain activation in response to same-as-previously- seen (OLD) vs. similar-to-previously-seen (SIM) objects in first episode psychosis (FEP) subjects before and after anti psychotic treatment and in matched healthy controls (HC). The current study uses three novel high-resolution task-based and post-encoding resting fMRI measures to probe hippocampal circuitry in delusions. It will also study CA1 function, using a sequential associative mismatch paradigm, as reflected by activation of CA1 in response to mismatching information compared to memory of that stimulus in FEP subjects before and after antipsychotic treatment and in matched HC. Finally, this study will evaluate plasticity of hippocampal intrinsic functional connectivity (IFC) in response to memory consolidation, using an encoding-plasticity paradigm, in FEP subjects before and after anti psychotic treatment and in matched HC. For each of the three imaging projects, a total of 50 FEP subjects and 50 matched healthy controls (HC) will be studied; hence, 300 subjects will be studied over 5 years. Within each paradigm, medication-naive FEP subjects will be studied at baseline and 8 weeks after starting anti psychotic medication. HC participants will be studied at baseline and 8 weeks later but will not receive any treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 16 to 35 years of age, inclusive, at the time of informed consent
* Right-handed
* Must have experienced a first episode of non-affective psychosis over the past five years
* Must exhibit a persistence of delusions for at least 4 days per week for at least 4 weeks in the absence of psychotomimetic substance use or other potential organic etiologies, including epilepsy or significant head trauma.
* Must score at least a 2 (mild to moderate) on the "Amount of preoccupation with delusions" and "Conviction" items on the Psychotic Symptom Rating Scale (PSYRATS).

Exclusion Criteria:

* Diagnosis of major mood disorder or other Axis I disorder other than Schizophrenia, Schizoaffective Disorder or Schizophreniform Disorder.
* Significant medical or neurological illness by history or physical exam including seizure disorder, history of loss of consciousness related to head trauma or developmental disorder including mental retardation.
* Metal implants, pacemaker, or other metal in the body or medicinal patch.
* History of claustrophobia.
* Currently taking any anti psychotic medication (within 4 weeks).

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Males and females with First Episode Psychosis
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2019-07-13 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
The difference in CA1 activation between a mismatch and an intact trial in FEP subjects after 8 weeks of antipsychotic treatment and the correlation of this change with change in delusions as measured by the Psyrats-D total score. | 8 Weeks
Change in hippocampus-to-VTA (hip-VTA) IFC and hip-to-lateral occipital complex (hip-LO) IFC, from pre- to post- encoding during the encoding-plasticity paradigm, between FEP and HC. | 8 Weeks
Change in (a) hip-VTA IFC and (b) hip-LO IFC, from pre- to post- encoding during the encoding-plasticity paradigm | 8 Weeks
correlation of change (a) hip-VTA IFC and (b) hip-LO IFC with change in delusional severity measured by the Psyrats-D total score. | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, MD, Principal Investigator — NYU Langone Health
Locations (3):
- New York Langone Health, New York, New York, United States
- China (2):
  - Shanghai Mental Health Center, Shanghai
  - Suzhou Guangji Hospital, Suzhou

IPD SHARING:
Plan to Share IPD: Yes
To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: All of the individual participant data collected during the trial, after deidentification.Researchers who provide a methodologically sound proposal will have access.